CLINICAL TRIAL: NCT06650059
Title: Cohort Study of Sickle Cell Patients Evaluating Analgesic Strategies and Their Consequences
Acronym: DDAM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240635; 2024-A01209-38 (Other: IDRCB number)
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease; Intense painful vaso-occlusive crises (VOC); Opioid use disorder (OUD)
MeSH Terms: conditions — Anemia, Sickle Cell; Opioid-Related Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Adult sickle cell patients followed in a sickle cell reference center (hôpital Henri Mondor, hôpital Necker-Enfants Malades and hôpital européen Georges-Pompidou, Assistance Publique-Hôpitaux de Paris).
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Self-questionnaire intended to each patient with sickle cell disease seen in consultation in one of the three reference centers participating in the study. Patients will complete the questionnaire once, on site.

SUMMARY:
To date, there is no comprehensive data among adults with sickle cell disease concerning the prevalence of consumption of level 2 and 3 analgesics at home and the use of cannabis or CBD for analgesic use. Preliminary data shows a very high prevalence of an opioid use disorder (OUD) in these patients, above 50%, but more precise additional studies are necessary to objectify these results and implement appropriate multidisciplinary care.

The general objective of this project is to establish an exhaustive collection on the addiction of sickle cell patients followed in a sickle cell reference center (hôpital Henri Mondor, hôpital Necker-Enfants Malades and hôpital européen Georges-Pompidou, Assistance Publique-Hôpitaux de Paris). The study investigative team proposes to set up a prospective observational study using a questionnaire.

DETAILED DESCRIPTION:
Sickle cell disease is one of the most common genetic diseases in the world with approximately 300,000 births per year of children with sickle cell disease. It is linked to the presence of a mutation on the beta globin chain (beta S mutation), responsible for the expression of the S variant of hemoglobin (HbS). Inherited autosomal recessively, is characterized, among other things, by intense painful vaso-occlusive crises (VOC) of bone triggered by cold, dehydration, stress or fatigue, but also sometimes without an identified triggering factor. The management of VOC requires, among other things, the rapid administration of analgesics. Level 1 seems ineffective and patients most often resort to level 2 from the start of symptoms, then level 3 in a hospital setting if the latter are ineffective. Sickle cell patients also frequently present with chronic pain, sometimes linked to complications of the disease (chronic leg ulcers, osteonecrosis in particular) but also without an identified cause.

The prescription of level 2 is therefore quite widely used in these patients for both the management of acute and chronic pain. In addition, self-management of pain has been encouraged for several years by caregivers, with the risk of more or less controlled self-medication, but little data is available in the literature.

Consequently, repeated exposure to opioids, as well as the painful context, constitute risk factors for the development of an opioid use disorder (OUD).

To date, there is no comprehensive data among adults with sickle cell disease concerning the prevalence of consumption of level 2 and 3 analgesics at home and the use of cannabis or CBD for analgesic use. Preliminary data shows a very high prevalence of OUD in these patients, above 50%, but more precise additional studies are necessary to objectify these results and implement appropriate multidisciplinary care.

The general objective of this project is to establish an exhaustive collection on the addiction of sickle cell patients followed in a sickle cell reference center (hôpital Henri Mondor, hôpital Necker-Enfants Malades and hôpital européen Georges-Pompidou, Assistance Publique-Hôpitaux de Paris). The study investigative team proposes to set up a prospective observational study using a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient.
* Sickle cell patient benefiting from a consultation or a session in a day hospital in one of the three reference centers (Necker Hospital, Mondor Hospital, Georges Pompidou European Hospital).
* Patient informed of the study and not opposed to participating in the research.

Exclusion Criteria:

* Patient under guardianship or curatorship.
* Non-literate patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult sickle cell patient cared in one of the three reference centers (Necker Hospital, Mondor Hospital, Georges Pompidou European Hospital).
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Diagnosis of opioid use disorder | Time 0
  The diagnosis of OUD will be established according to the criteria of the 5th version of the Diagnostic and Statistical Manual of Mental Illnesses (DSM 5). In this version the diagnosis of a use disorder is made if a patient meets 2 criteria among the 11 specified over a period of at least 12 months. These criteria cover four dimensions: loss of control over consumption (4 criteria), social impairment of functioning (3 criteria), continuation of use despite the risks incurred or presented (2 criteria), and physical symptoms (2 criteria). Depending on the number of criteria met, a gradation of severity is established: mild OUD (2 to 3 criteria), moderate (4 to 5 criteria), or severe (6 criteria or more).

SECONDARY OUTCOMES:
Cannabis use | Time 0
  Current and past cannabis consumption will be assessed by a closed question. As for problematic use, it will be sought using the CAST questionnaire (Cannabis Abuse Screening Test), a 6-item scale that describes the behavior of use or problems experienced within the scope of cannabis use. Each of these items describes usage behaviors or problems encountered in the context of cannabis consumption:on use in the morning or alone, that is to say assumed outside of a festive context; possible disorders of the memory; being encouraged to reduce or stop drinking; failures in attempts to stop; problems such as fights, accidents, etc. following consumption of cannabis. The effects felt after taking cannabis will also be researched. To calculate the score, the modalities are coded from 0 to 4. The total obtained vary from 0 to 24.A risk-free users is defined when they have a score less than 3, the users with a low risk for a score = 3 and <7 and a high risk dependency for a score = or ˃7.
Consumption of CBD for analgesic purposes | Time 0
  CBD consumption for analgesic purposes will be assessed by a closed question.
Tobacco consumption | Time 0
  The existence of tobacco consumption will be assessed by a closed question on current and lifetime smoking. The severity of dependence will be assessed by the Fagerström questionnaire. It includes 10 questions relating to the smoker's consumption habits. Depending on the answers given, a score of 0 to 10 is obtained; dependence is thus judged to be zero if the score is 0 to 2, weak 3 or 4, average 5 or 6, strong 7 or 8 and very strong 9 or 10.
Use of vaping | Time 0
  The use of vaping will be assessed by a closed question.
Factors linked to sickle cell disease and associated with substance use: opioids, cannabis, CBD and tobacco | Time 0
  The factors linked to sickle cell disease and associated with the use of substances: opioids, cannabis, CBD and tobacco, will be collected by closed questions and are :
  * Patient characteristics: sex, country, month and year of birth, marital status, professional activity,
  * History of sickle cell disease: description and evolution of vaso-occlusive crises (VOC), chronic pain, and complications,
  * Current therapies: current drug treatments, use of analgesics during the last 12 months, and other non-drug therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Laure Joseph, M.D., Principal Investigator — Assistance Publique - Hôpitaux de Paris; Elena Foïs, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Hôpital Henri Mondor, Créteil
  - Hôpital européen Georges-Pompidou, Paris
  - Hôpital Necker-Enfants Malades, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elander J, Lusher J, Bevan D, Telfer P, Burton B. Understanding the causes of problematic pain management in sickle cell disease: evidence that pseudoaddiction plays a more important role than genuine analgesic dependence. J Pain Symptom Manage. 2004 Feb;27(2):156-69. doi: 10.1016/j.jpainsymman.2003.12.001. PMID 15157040
- [Background] Feliu MH, Wellington C, Crawford RD, Wood M, Edwards L, Byrd G, Edwards CL. Opioid management and dependency among adult patients with sickle cell disease. Hemoglobin. 2011;35(5-6):485-94. doi: 10.3109/03630269.2011.610914. Epub 2011 Sep 12. PMID 21910605
- [Background] Al Zahrani O, Hanafy E, Mukhtar O, Sanad A, Yassin W. Outcomes of multidisciplinary team interventions in the management of sickle cell disease patients with opioid use disorders. A retrospective cohort study. Saudi Med J. 2020 Oct;41(10):1104-1110. doi: 10.15537/smj.2020.10.25386. PMID 33026052
- [Background] Gerardin M, Couec ML, Grall-Bronnec M, Feuillet F, Wainstein L, Rousselet M, Pinot ML, Perrouin F, Bonnot O, Drouineau MH, Jolliet P, Victorri-Vigneau C. PHEDRE trial protocol - observational study of the prevalence of problematic use of Equimolar Mixture of Oxygen and Nitrous Oxide (EMONO) and analgesics in the French sickle-cell disease population. BMC Psychiatry. 2015 Nov 14;15:281. doi: 10.1186/s12888-015-0677-5. PMID 26573686
- [Background] Abrams DI, Couey P, Dixit N, Sagi V, Hagar W, Vichinsky E, Kelly ME, Connett JE, Gupta K. Effect of Inhaled Cannabis for Pain in Adults With Sickle Cell Disease: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jul 1;3(7):e2010874. doi: 10.1001/jamanetworkopen.2020.10874. PMID 32678452
- [Background] Gerardin M, Rousselet M, Couec ML, Masseau A, Guerlais M, Authier N, Deheul S, Roussin A, Micallef J, Djezzar S; French Addictovigilance Network (FAN); Feuillet F, Jolliet P, Victorri-Vigneau C. Descriptive analysis of sickle cell patients living in France: The PHEDRE cross-sectional study. PLoS One. 2021 Mar 18;16(3):e0248649. doi: 10.1371/journal.pone.0248649. eCollection 2021. PMID 33735176